CLINICAL TRIAL: NCT05581641
Title: An Exploratory Phase I, Randomized, Observer-blind, Placebo-controlled Dose Escalation Trial Evaluating the Safety, Tolerability and Immunogenicity of an Investigational RNA-based Vaccine for Active Immunization Against Malaria
Brief Title: Safety and Immune Responses After Vaccination With an Investigational RNA-based Vaccine Against Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: BNT165-01
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Malaria
Keywords: RNA vaccine; Vaccine; Active immunization against malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: observer-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: BNT165b1: 3 Micrograms (mcg) (Experimental): Participants received 3 intramuscular injections of 3 mcg of BNT165b1 vaccine, one each at Days 1, 57 and 183, respectively.
  Interventions: Biological: BNT165b1
- Cohort 2: BNT165b1: 10 mcg (Experimental): Participants received 3 intramuscular injections of 10 mcg of BNT165b1 vaccine, one each at Days 1, 57 and 183, respectively.
  Interventions: Biological: BNT165b1
- Cohort 3: BNT165b1: 30 mcg (Experimental): Participants received 3 intramuscular injections of 30 mcg of BNT165b1 vaccine, one each at Days 1, 57 and 183, respectively.
  Interventions: Biological: BNT165b1
- Placebo (Placebo Comparator): Participants received 3 intramuscular injections of matching placebo of BNT165b vaccine, one each at Days 1, 57 and 183, respectively.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT165b1 — RNA vaccine for active immunization against malaria administered as intramuscular injection.
  Arms: Cohort 1: BNT165b1: 3 Micrograms (mcg); Cohort 2: BNT165b1: 10 mcg; Cohort 3: BNT165b1: 30 mcg
Other: Placebo — Placebo matched to RNA vaccine administered as intramuscular injection.
  Arms: Placebo

SUMMARY:
This first-in-human clinical trial, was a dose escalation multi-center trial designed to assess the safety, tolerability, and immunogenicity of the vaccine component, BNT165b1, a ribonucleic acid (RNA)-lipid nanoparticle (LNP) encoding for part of the Plasmodium falciparum circumsporozoite protein (PfCSP).

BNT165b1 was evaluated at three dose levels (DLs) to select a safe and tolerable dose in a 3-dose schedule.

DETAILED DESCRIPTION:
The trial had enrolled participants into three cohorts by dose level who were randomized 4:1 to BNT165b1: placebo. The trial used a staggered dose escalation schema with sentinel participants for Dose 1 in all cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Had given informed consent by signing and dating the informed consent form (ICF) before initiation of any trial-specific procedures
* Were willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions (e.g., to follow good practices to reduce their chances of being infected or spreading Coronavirus Disease 2019 [COVID-19]), and other requirements of the trial. This includes that they were able to understand and follow trial-related instructions
* Were aged 18 to 55 years, had a body mass index over 18.5 kg/m^2 and under 35 kg/m^2 and weighed at least 45 kg at Visit 0
* Were healthy, in the clinical judgment of the investigator based on volunteer-reported medical history data, and physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory test outcomes at Visit 0

  * Note: Healthy volunteers with pre-existing stable disease (e.g., obesity, hypertension), defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 90 days before Visit 0, were included
* Agreed not to enroll in another trial with an investigational medicinal product (IMP) starting from Visit 0 and until 12 weeks after receiving Dose 3
* Agreed not to travel to a malaria endemic region starting from Visit 0 and until 28 days after Dose 3, as defined per CDC (Centers for Disease Control and Prevention)
* Negative human immunodeficiency virus (HIV) -1 and -2 blood test result at Visit 0
* Negative severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) antigen test result at Visit 0
* Negative hepatitis B surface antigen (HBsAg) test result at Visit 0 and negative anti Hepatitis C virus (anti-HCV) antibodies, or negative HCV polymerase chain reaction test result if the anti-HCV was positive at Visit 0
* Volunteers of childbearing potential (VOCBP) who had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test result at Visit 0 and negative urine pregnancy test results before each IMP administration. Volunteers born female who were postmenopausal or permanently sterilized were not considered VOBCP
* VOCBP who agreed to practice a highly effective form of contraception and required their male sexual partners to use condoms with a spermicidal agent, starting at Visit 0 and continuously until 90 days after receiving Dose 3
* VOCBP who agreed not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting at Visit 0 and continuously until 90 days after receiving Dose 3
* Men who were sexually active with partners of childbearing potential and who did not have a vasectomy that agreed to use condoms with a spermicidal agent and to practice a highly effective form of contraception with their sexual partners born female during the trial, starting at Visit 0 and continuously until 90 days after receiving Dose 3
* Men who were willing to refrain from sperm donation, starting at Visit 0 and continuously until 90 days after receiving Dose 3

Exclusion Criteria:

* History of malaria infection (any species) based on volunteer-reported medical history
* Travel to a malaria endemic region starting 6 months before Visit 0 and continuously until 28 days after receiving Dose 3, as defined per CDC
* Prior residence for greater than or equal to (>=) 6 months in a malaria endemic region
* Were breastfeeding or had intended to become pregnant starting with Visit 0 and continuously until 90 days after receiving Dose 3 or fathered children starting with Visit 0 and continuously until 90 days after receiving Dose 3
* History of any serious adverse reactions to vaccines or to vaccine components such as lipids and including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had an anaphylactic adverse reaction to pertussis vaccine as a child).
* Current or history of the following medical conditions:

  1. Uncontrolled or moderate or severe respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease); symptoms of asthma severity as defined in the US National Asthma Education and Prevention Program Expert Panel report, 2020 - e.g., exclude a volunteer who:

     * Used a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
     * Used high dose inhaled corticosteroids (per American Academy of Allergy Asthma & Immunology), or
     * In the past year has had either of the following:

       * Greater than one exacerbation of symptoms treated with oral/parenteral corticosteroids;
       * Needed hospitalization, or intubation for asthma.
  2. Diabetes mellitus type 1 or type 2, including cases controlled with diet alone (Not excluded: history of isolated gestational diabetes).
  3. Hypertension:

     * If a person had been found to have elevated blood pressure or hypertension during screening or previously, they were excluded for blood pressure that is not well controlled. Well controlled blood pressure was defined as consistently less than or equal to (<=)140 mm Hg systolic and <= 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be <= 150 mm Hg systolic and <=100 mm Hg diastolic at enrollment.
     * If a person did not have a history of elevated blood pressure or hypertension previously or during screening, also excluded for systolic blood pressure greater than (>)150 mm Hg at enrollment or diastolic blood pressure ≥100 mm Hg at enrollment.
  4. Malignancy within 5 years of screening, excluding localized basal or squamous cell cancer;
  5. Any current or history of cardiovascular diseases, (e.g., myocarditis, pericarditis, myocardial infarction, congestive heart failure, cardiomyopathy or clinically significant arrhythmias), unless such disease was not considered relevant for participation in this trial in the investigator's judgment;
  6. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions);
  7. Seizure disorder: History of seizure(s) within past 3 years. Also excluded if volunteer had used medications in order to prevent or treat seizure(s) at any time within the past 3 years
* Documented major psychiatric illness, including bipolar disorder, major depressive disorder, schizophrenia, autism, and attention deficit-hyperactivity disorder that at the discretion of the investigator could interfere with participation and follow-up as outlined by the trial
* The following diseases associated with immune dysregulation:

  * Primary immunodeficiencies.
  * History of solid organ or bone marrow transplantation.
  * Asplenia: any condition resulting in the absence of a functional spleen.
  * Currently existing or history of autoimmune disease including and not limited to thyroid autoimmune disease, multiple sclerosis, psoriasis, etc.
* Previous vaccination with an approved or investigational malaria vaccine at any time or having taken part in a human malaria challenge study
* Receipt of any investigational product within 28 days before Visit 0
* Any planned non-trial vaccinations starting at Visit 0 and continuously until Visit 11 (28 days after Dose 3)

  * Note: Seasonal influenza and COVID-19 vaccines were allowed; however, they should have been administered at least 14 days before or after any IMP injection
* Received blood/plasma products or immunoglobulin within 120 days before Visit 1 or planned administration starting at Visit 0 and continuously until Visit 12
* Received allergy treatment with antigen injections within 28 days before first IMP administration or that were scheduled within 14 days after Visits 1, 5 and 9
* Current or planned treatment with immunosuppressive therapy, including systemic corticosteroids (if systemic corticosteroids are administered for >=14 days at a dose of >= 20 mg/day of prednisone or equivalent) starting at Visit 0 and continuously until Visit 11 (28 days after Dose 3). Intraarticular, intrabursal, or topical (skin or eyes) corticosteroids were permitted
* Had a history of alcohol abuse or drug addiction within 1 year before Visit 0 or had a history (within the past 5 years) of substance abuse which in the opinion of the investigator, could compromise their wellbeing if they participate as participants in the trial, or that could prevent, limit, or confound the protocol-specified assessments
* Any existing condition which may have affected vaccine injection and/or assessment of local reactions assessment at the injection site, e.g., tattoos, severe scars, etc.
* Were vulnerable individuals as per International Council for Harmonization (ICH) E6 definition, i.e., were individuals whose willingness to volunteer in a clinical trial may have been unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate
* Any screening hematology and/or blood chemistry laboratory value that met the definition of a Grade >= 2 abnormality or of Grade 1 at the investigator's discretion at Visit 0. Individuals with abnormal but not clinically significant parameters were not included in the toxicity guidance may have been considered eligible at the discretion of the investigator
* Had current febrile illness (body temperature >=38.0°C/ >=100.4°F) or febrile illness within 48 hours of Visit 0

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (5):
- United States (5):
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - University of Maryland, Center for Vaccine Development, Baltimore, Maryland
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mo AX, McGugan G, Pesce JT. Meeting report: Expert consultation on late arresting replication competent (LARC) malaria sporozoite vaccine research & development. Vaccine. 2025 Apr 30;54:127009. doi: 10.1016/j.vaccine.2025.127009. Epub 2025 Apr 16. PMID 40245769

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: BNT165b1: 3 Micrograms (mcg) | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
Started | 16 | 16 | 16 | 12
Vaccinated With Dose 1 (Day 1) | 16 | 16 | 16 | 12
Vaccinated With Dose 2 (Day 57) | 15 | 15 | 14 | 10
Vaccinated With Dose 3 (Day 183) | 15 | 15 | 13 | 9
Completed | 14 | 14 | 11 | 9
Not Completed | 2 | 2 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the safety set that included all participants who received at least one dose of the investigational medicinal product (IMP).
Groups:
- Cohort 1: BNT165b1: 3 mcg: Participants received 3 intramuscular injections of 3 mcg of BNT165b1 vaccine, one each at Days 1, 57 and 183, respectively.
- Placebo: Participants received 3 intramuscular injections of matching placebo of BNT165b1 vaccine, one each at Days 1, 57 and 183, respectively.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.61) | 41.5 (10.46) | 35.6 (10.14) | 34.2 (10.16) | 38.8 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 4 | 6 | 30
  Male | 5 | 7 | 12 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 6 | 1 | 15
  Not Hispanic or Latino | 16 | 8 | 10 | 11 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 2 | 2 | 4 | 10
  White | 14 | 14 | 12 | 7 | 47
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter square (kg/m^2)] | 28.05 (3.665) | 28.85 (3.195) | 26.06 (3.954) | 27.28 (4.564) | 27.58 (3.875)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Reactions
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) and pre-listed (that is, solicited) in the e-diary. Solicited local reactions included: pain at the injection site, erythema/redness, and induration/swelling. The intensity of AEs was graded by the investigator. Grades were defined as: Grade 1 - Mild; does not interfere with the trial participant's usual function; Grade 2 - Moderate; interferes to some extent with the trial participant's usual function; Grade 3 - Severe; interferes significantly with the trial participant's usual function and Grade 4 - Potentially life-threatening; life-threatening consequences, urgent intervention required. Participants may have been counted more than once if they reported multiple episodes of the event for the specified doses.
Time Frame: Up to 7 days post any vaccination, and up to 7 days post each vaccination dose (i.e., post Dose 1 [at Day 8], Dose 2 [at Day 64] and Dose 3 [at Day 190])
Population: Analysis was performed on the safety set, i.e., participants who received at least one dose of the IMP. Here, "number analyzed" signified participants who received vaccination at the specified visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 12
Participants
  Erythema/Redness- Post any vaccination | 0 | 1 | 1 | 0
  Induration/Swelling- Post any vaccination | 0 | 2 | 0 | 0
  Pain at the injection site- Post any vaccination | 4 | 6 | 9 | 1
  Erythema/Redness- Post Dose 1 | 0 | 0 | 0 | 0
  Induration/Swelling- Post Dose 1 | 0 | 1 | 0 | 0
  Pain at the injection site- Post Dose 1 | 2 | 4 | 8 | 0
  Erythema/Redness- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Erythema/Redness- Post Dose 2 | 0 | 0 | 0 | 0
  Induration/Swelling- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Induration/Swelling- Post Dose 2 | 0 | 0 | 0 | 0
  Pain at the injection site- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Pain at the injection site- Post Dose 2 | 2 | 3 | 5 | 1
  Erythema/Redness- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Erythema/Redness- Post Dose 3 | 0 | 1 | 1 | 0
  Induration/Swelling- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Induration/Swelling- Post Dose 3 | 0 | 1 | 0 | 0
  Pain at the injection site- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Pain at the injection site- Post Dose 3 | 3 | 4 | 5 | 0
  Grade >=3 Local Reaction-Post Dose 1 | 0 | 0 | 0 | 0
  Grade >=3 Local Reaction-Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Grade >=3 Local Reaction-Post Dose 2 | 0 | 0 | 0 | 0
  Grade >=3 Local Reaction-Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Grade >=3 Local Reaction-Post Dose 3 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) pre-listed (i.e., solicited) in the e-diary. Solicited systemic reactions included: vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, and fever. The intensity of AEs was graded by the investigator. Grades were defined as: Grade 1 - Mild; does not interfere with the trial participant's usual function; Grade 2 - Moderate; interferes to some extent with the trial participant's usual function; Grade 3 - Severe; interferes significantly with the trial participant's usual function and Grade 4 - Potentially life-threatening; life-threatening consequences, urgent intervention required. Participants may have been counted more than once if they reported multiple episodes of the event for the specified doses.
Time Frame: as for outcome 1
Population: Analysis was performed on the safety set. Here, "number analyzed" signified participants who received vaccination at the specified visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 12
Participants
  Arthralgia- Post any vaccination | 2 | 3 | 1 | 1
  Chills- Post any vaccination | 1 | 4 | 0 | 1
  Diarrhea- Post any vaccination | 5 | 3 | 2 | 1
  Fatigue- Post any vaccination | 9 | 8 | 5 | 4
  Fever- Post any vaccination | 0 | 0 | 0 | 0
  Headache- Post any vaccination | 6 | 8 | 5 | 2
  Myalgia- Post any vaccination | 4 | 5 | 4 | 2
  Vomiting- Post any vaccination | 1 | 0 | 1 | 0
  Arthralgia- Post Dose 1 | 0 | 2 | 1 | 1
  Chills- Post Dose 1 | 1 | 3 | 0 | 0
  Diarrhea- Post Dose 1 | 2 | 3 | 1 | 1
  Fatigue- Post Dose 1 | 7 | 8 | 3 | 3
  Fever- Post Dose 1 | 0 | 0 | 0 | 0
  Headache- Post Dose 1 | 4 | 5 | 2 | 1
  Myalgia- Post Dose 1 | 1 | 3 | 3 | 1
  Vomiting- Post Dose 1 | 1 | 0 | 1 | 0
  Arthralgia- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Arthralgia- Post Dose 2 | 1 | 1 | 0 | 0
  Chills- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Chills- Post Dose 2 | 0 | 0 | 0 | 0
  Diarrhea-Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Diarrhea-Post Dose 2 | 3 | 0 | 1 | 0
  Fatigue- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Fatigue- Post Dose 2 | 3 | 2 | 3 | 2
  Fever- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Fever- Post Dose 2 | 0 | 0 | 0 | 0
  Headache- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Headache- Post Dose 2 | 1 | 1 | 3 | 0
  Myalgia- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Myalgia- Post Dose 2 | 2 | 3 | 1 | 1
  Vomiting- Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Vomiting- Post Dose 2 | 0 | 0 | 0 | 0
  Arthralgia- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Arthralgia- Post Dose 3 | 1 | 0 | 0 | 1
  Chills- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Chills- Post Dose 3 | 0 | 1 | 0 | 1
  Diarrhea- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Diarrhea- Post Dose 3 | 1 | 0 | 0 | 0
  Fatigue- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Fatigue- Post Dose 3 | 1 | 3 | 3 | 2
  Fever- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Fever- Post Dose 3 | 0 | 0 | 0 | 0
  Headache- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Headache- Post Dose 3 | 3 | 2 | 1 | 2
  Myalgia- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Myalgia- Post Dose 3 | 2 | 0 | 0 | 2
  Vomiting- Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Vomiting- Post Dose 3 | 0 | 0 | 0 | 0
  Grade >=3 Systemic Reaction-Post Dose 1 | 0 | 0 | 0 | 0
  Grade >=3 Systemic Reaction-Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Grade >=3 Systemic Reaction-Post Dose 2 | 0 | 0 | 0 | 0
  Grade >=3 Systemic Reaction-Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Grade >=3 Systemic Reaction-Post Dose 3 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered with a pharmaceutical product, and which did not necessarily have a causal relationship with this treatment. The intensity of AEs was graded by the investigator. Grades were defined as: Grade 1 - Mild; does not interfere with the trial participant's usual function; Grade 2 - Moderate; interferes to some extent with the trial participant's usual function; Grade 3 - Severe; interferes significantly with the trial participant's usual function and Grade 4 - Potentially life-threatening; life-threatening consequences, urgent intervention required. Participants may have been counted more than once if they reported multiple episodes of the event for the different doses.
Time Frame: Up to 28 days post any vaccination, and up to 28 days post each vaccination dose (i.e., post Dose 1 [at Day 29], Dose 2 [at Day 85] and Dose 3 [at Day 211])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 12
Participants
  Post any vaccination | 4 | 7 | 4 | 3
  Post Dose 1 | 1 | 4 | 3 | 1
  Any Grade >= 3 AE: Post Dose 1 | 0 | 0 | 1 | 0
  Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Post Dose 2 | 3 | 1 | 1 | 1
  Any Grade >= 3 AE: Post Dose 2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Any Grade >= 3 AE: Post Dose 2 | 0 | 0 | 0 | 0
  Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Post Dose 3 | 0 | 2 | 2 | 2
  Any Grade >= 3 AE: Post Dose 3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Any Grade >= 3 AE: Post Dose 3 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death and was life-threatening. It also included any event requiring hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, caused a congenital anomaly or birth defect, or any other event determined as SAE as per medical or scientific judgment.
Time Frame: From Day 1 up to 24 weeks after Dose 3 (i.e., up to Day 351)
Population: Analysis was performed on the safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 12
Participants | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs)
Description: MAAE was defined as an AE for which the participants received medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits. Participants may have been counted more than once if they reported multiple episodes of the event for the different doses.
Time Frame: Up to 28 days post any vaccination, and up to 28 days post each vaccination dose (i.e., post Dose 1 [at Day 29], Dose 2 [at Day 85], Dose 3 [at Day 211])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 12
Participants
  Post any vaccination | 2 | 3 | 2 | 1
  Post Dose-1 | 0 | 0 | 1 | 0
  Post Dose-2: number analyzed (Participants) | 15 | 15 | 14 | 10
  Post Dose-2 | 2 | 1 | 1 | 0
  Post Dose-3: number analyzed (Participants) | 15 | 15 | 13 | 9
  Post Dose-3 | 0 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: AE data were collected from Day 1 up to 28 days after each vaccination. All SAEs collected throughout the study are reported in the AE section and were reported from Visit 0 (Screening) up to Visit 14 (i.e., 1 year post Dose 3, up to Day 548)
Description: Analysis was performed on the safety set. Per protocol, solicited local and systemic reactions were not included in the AE analysis unless they continued longer than 7 days post-investigational medicinal product (IMP) administration or were a SAE. Solicited local and systemic reactions are presented in the respective outcome measures.
Arm/Group | Cohort 1: BNT165b1: 3 mcg | Cohort 2: BNT165b1: 10 mcg | Cohort 3: BNT165b1: 30 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 4/16 | 7/16 | 4/16 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BNT165b1: 3 mcg (N=16) | Cohort 2: BNT165b1: 10 mcg (N=16) | Cohort 3: BNT165b1: 30 mcg (N=16) | Placebo (N=12)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BNT165b1: 3 mcg (N=16) | Cohort 2: BNT165b1: 10 mcg (N=16) | Cohort 3: BNT165b1: 30 mcg (N=16) | Placebo (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — Includes also solicited systemic reactions that continued longer than 7 days post-IMP administration.
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 1 — Includes also solicited systemic reactions that continued longer than 7 days post-IMP administration.
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 2
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 — Includes also solicited systemic reactions that continued longer than 7 days post-IMP administration.
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Includes also solicited systemic reactions that continued longer than 7 days post-IMP administration.
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 — Includes also solicited systemic reactions that continued longer than 7 days post-IMP administration.
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT05581641/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT05581641/SAP_001.pdf